CLINICAL TRIAL: NCT03935438
Title: The Influence of Cardiac Rehabilitation on the Health State of Patients After Acute Coronary Syndrome
Brief Title: The Influence of Cardiac Rehabilitation on the Health State After ACS
Acronym: CARDIO-REH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Damian Skrypnik, Principal Investigator and Study Manager; Doctor of Medicine, Poznan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 476/19
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Rehabilitation; Acute Coronary Syndrome
Keywords: cardiac rehabilitation; acute coronary syndrome; anthropometric parameters; physical efficiency; cardiovascular function
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients after ACS (Experimental): Patients after acute coronary syndrome undergoing cardiac rehabilitation.
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation — The training program of cardiac rehabilitation, depending on the results of the patient's medical qualification, will consist of the following: free active exercises, isometric exercises, active exercises in relief with resistance, isotonic exercises, isokinetic exercises, active breathing exercises, active breathing exercises with resistance, balance exercises, general exercises- individual and in groups, interval training on a treadmill or cycling cycloergometer, continuous training on a treadmill or cycling cycloergometer, circuit training, walking training, march training with accessories, autogenic training, walking. The training program will last an average 2 weeks.

SUMMARY:
Coronary heart disease, including acute coronary syndromes (ACS), is the leading cause of death in European countries. One of the basic elements of secondary and tertiary prevention of ACS is cardiac rehabilitation.

The aims of the study are evaluation of the impact of cardiac rehabilitation on health state- especially on cardiovascular function parameters in patients after acute coronary syndrome and evaluation of the influence of the level of gene expression and polymorphisms of genes associated with ischemic heart disease on the course of cardiac rehabilitation in patients after ACS.

The study will consist of a retrospective and prospective part. The retrospective part will include patients who have had acute coronary syndrome in the past and then - before being included in the study - have undergone cardiac rehabilitation. In the retrospective part, patients enrolled in the study will not undergo cardiac rehabilitation as a part of the study intervention. The prospective part will include patients who have had an acute coronary syndrome in the past and will undergo cardiac rehabilitation as the study intervention.

After being included in the study, patients will undergo medical examination. Then subsequent procedures will be performed: anthropometric measurements; ECG; body composition analysis by bioimpedance; measurement of resting blood pressure, resting heart rate and oxygen saturation of hemoglobin; pulse wave analysis; transthoracic echocardiography of the heart; 24-hour blood pressure measurement by ambulatory blood pressure monitoring (ABPM); 24-hour ECG recording using the Holter method; electrocardiographic exercise test on a treadmill and / or a six-minute walk test or other exercise test adequate to the patient's state of health; assessment of the quality of the diet; assessment of lifestyle, acceptance of disease and quality of life; assessment of the psychological profile.

Subsequently patients taking part in the prospective part of the study will perform a cardiac rehabilitation program.

After the cardiac rehabilitation program measurement procedures listed above will be repeated.

Before and after the cardiac rehabilitation program blood samples, urine samples and hair samples will be collected. Blood samples, urine samples and hair samples will also be collected from patients taking part in the retrospective part of the study.

DETAILED DESCRIPTION:
Coronary heart disease, including acute coronary syndromes (ACS), is the leading cause of death in European countries, including Poland. In addition, it is one of the main causes of disability and the number of lost years of life and the number of years of life lost in good health. The costs of its treatment include not only the primary prophylaxis of cardiovascular events, the treatment of cardiovascular events, the treatment of chronic conditions and complications such as chronic heart failure or arrhythmia, but also the secondary and tertiary prophylaxis of acute coronary syndromes.

One of the basic elements of secondary and tertiary prevention of ACS is cardiac rehabilitation. It should be implemented as soon as possible after the ACS and be part of a comprehensive, planned and systematic care of the patient after ACS. The beneficial effect of cardiac rehabilitation on the cardiovascular system, lipid and carbohydrate metabolism and physical performance has been demonstrated in a way that does not raise any doubts. However, in the light of the growing epidemic of civilization diseases such as excessive body mass, diabetes, dyslipidemia, hypertension and other cardiometabolic disorders, it is necessary to conduct high-quality research on the development of the most effective cardiac rehabilitation programs, so as to maximize their beneficial effect on patients' health.

The aims of the study are:

1. Evaluation of the impact of cardiac rehabilitation on selected anthropometric, biochemical, mineral parameters, body composition parameters, physical fitness parameters and cardiovascular function parameters in patients after acute coronary syndrome.
2. Assessment of lifestyle, acceptance of disease, quality of life, diet and psychological profile and the influence of these factors on the course of cardiac rehabilitation in patients after acute coronary syndrome.
3. Evaluation of the influence of the level of gene expression and polymorphisms of genes associated with ischemic heart disease and predisposing conditions (including excessive body weight, hypertension, lipid and carbohydrate disorders, impaired vascular endothelial function) on the course of cardiac rehabilitation in patients after acute coronary syndrome and searching for new genes that may affect the course of cardiac rehabilitation in this group of patients.

Research hypotheses:

1. Cardiac rehabilitation has a positive effect on selected anthropometric, biochemical, mineral parameters, body composition parameters, physical fitness parameters and cardiovascular function parameters in patients after acute coronary syndrome.
2. Lifestyle, acceptance of disease, quality of life, diet and psychological profile have a significant impact on the course of cardiac rehabilitation in patients after acute coronary syndrome.
3. The level of expression and gene polymorphism of genes associated with ischemic heart disease and predisposing conditions (including excessive body weight, hypertension, lipid and carbohydrate disorders, impaired vascular endothelial function) have a significant impact on the course of cardiac rehabilitation in patients after acute coronary syndrome.

The study will consist of a retrospective and prospective part. The retrospective part will include patients who have had acute coronary syndrome in the past and then - before being included in the study - have undergone cardiac rehabilitation. In the retrospective part, patients enrolled in the study will not undergo cardiac rehabilitation as a part of the study intervention. In contrast, the prospective part will include patients who have had an acute coronary syndrome in the past and will undergo cardiac rehabilitation as the study intervention.

About 200 women and men aged 18 to 99 are planned to be included in the study.

After being included in the study, patients will undergo medical examination and their medical documentation will be collected, analyzed, copied and archived. Then subsequent procedures will be performed:

* anthropometric measurements (body weight, height, hip, waist, neck circumference measurement)
* ECG - electrocardiography
* non-invasive analysis of the body composition by bioimpedance
* non-invasive measurement of resting blood pressure, resting heart rate and oxygen saturation of hemoglobin
* non-invasive pulse wave analysis
* non-invasive transthoracic echocardiography of the heart
* non-invasive 24-hour blood pressure measurement by ABPM
* non-invasive 24-hour ECG recording using the Holter method
* non-invasive electrocardiographic exercise test on a treadmill and / or a six-minute walk test or other exercise test adequate to the patient's state of health; these tests will always be preceded by a detailed medical qualification
* assessment of the quality of the diet
* assessment of lifestyle, acceptance of disease and quality of life
* assessment of the psychological profile

Subsequently patients taking part in the prospective part of the study will perform a cardiac rehabilitation program.

After the cardiac rehabilitation program measurement procedures listed above (anthropometric measurements; ECG; non-invasive analysis of the body composition by bioimpedance; non-invasive measurement of resting blood pressure, resting heart rate and oxygen saturation of hemoglobin; non-invasive pulse wave analysis; non-invasive transthoracic echocardiography of the heart; non-invasive 24-hour blood pressure measurement by ABPM; non-invasive 24-hour ECG recording using the Holter method; non-invasive electrocardiographic exercise test; assessment of the quality of the diet; assessment of lifestyle, acceptance of disease and quality of life; assessment of the psychological profile) will be repeated.

Before and after the cardiac rehabilitation program blood samples, urine samples and hair samples will be collected. Blood samples, urine samples and hair samples will also be collected from patients taking part in the retrospective part of the study.

After data collection statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent in writing
* Coronary heart disease, a state after an acute coronary syndrome
* Female or male
* Age 18 - 99 years

Exclusion Criteria:

* Active neoplastic disease
* Alcohol abuse, drug abuse
* Pregnancy, lactation
* Other conditions that in the opinion of researchers may pose any risk to the patient during the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity (PWV) I | At baseline
  Pulse wave velocity I
PWV II | After intervention completion- an average of 2 weeks from baseline
  Pulse wave velocity II

SECONDARY OUTCOMES:
Aortic pressure (AP) I | At baseline
  Aortic pressure I
AP II | After intervention completion- an average of 2 weeks from baseline
  Aortic pressure II
Body mass (BM) I | At baseline
  Body mass I
BM II | After intervention completion- an average of 2 weeks from baseline
  Body mass II
Body height (BH) I | At baseline
  Body height I
BH II | After intervention completion- an average of 2 weeks from baseline
  Body height II
Body mass index (BMI) I | At baseline
  Body mass index I
BMI II | After intervention completion- an average of 2 weeks from baseline
  Body mass index II
Waist circumference (WC) I | At baseline
  Waist circumference I
WC II | After intervention completion- an average of 2 weeks from baseline
  Waist circumference II
Hip circumference (HC) I | At baseline
  Hip circumference I
HC II | After intervention completion- an average of 2 weeks from baseline
  Hip circumference II
Neck circumference (NC) I | At baseline
  Neck circumference I
NC II | After intervention completion- an average of 2 weeks from baseline
  Neck circumference II
Total fat percentage (TF%) I | At baseline
  Total fat percentage I
TF% II | After intervention completion- an average of 2 weeks from baseline
  Total fat percentage II
Systolic blood pressure (SBP) I | At baseline
  Systolic blood pressure I
SBP II | After intervention completion- an average of 2 weeks from baseline
  Systolic blood pressure II
Diastolic blood pressure (DBP) I | At baseline
  Diastolic blood pressure I
DBP II | After intervention completion- an average of 2 weeks from baseline
  Diastolic blood pressure II
Heart rate (HR) I | At baseline
  Heart rate I
HR II | After intervention completion- an average of 2 weeks from baseline
  Heart rate II
Blood oxygen saturation (SO2) I | At baseline
  Blood oxygen saturation I
SO2 II | After intervention completion- an average of 2 weeks from baseline
  Blood oxygen saturation II
Ejection fraction (EF) I | At baseline
  Ejection fraction I
EF II | After intervention completion- an average of 2 weeks from baseline
  Ejection fraction II
Ambulatory blood pressure monitoring- systolic blood pressure (ABPM SBP) I | At baseline
  Ambulatory blood pressure monitoring- systolic blood pressure I
ABPM SBP II | After intervention completion- an average of 2 weeks from baseline
  Ambulatory blood pressure monitoring- systolic blood pressure II
Ambulatory blood pressure monitoring- diastolic blood pressure (ABPM DBP) I | At baseline
  Ambulatory blood pressure monitoring- diastolic blood pressure I
ABPM DBP II | After intervention completion- an average of 2 weeks from baseline
  Ambulatory blood pressure monitoring- diastolic blood pressure II
Metabolic equivalent (MET) I | At baseline
  Metabolic equivalent I
MET II | After intervention completion- an average of 2 weeks from baseline
  Metabolic equivalent II
Distance in 6-minutes walk (6MW-D) I | At baseline
  Distance in 6-minutes walk I
6MW-D II | After intervention completion- an average of 2 weeks from baseline
  Distance in 6-minutes walk II
aspartate aminotransferase (AST) I | At baseline
  Blood concentration of aspartate aminotransferase I
AST II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of aspartate aminotransferase II
alanine aminotransferase (ALT) I | At baseline
  Blood concentration of alanine aminotransferase I
ALT II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of alanine aminotransferase II
total bilirubin (TB) I | At baseline
  Blood concentration of total bilirubin I
TB II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of total bilirubin II
indirect bilirubin (IB) I | At baseline
  Blood concentration of indirect bilirubin I
IB II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of indirect bilirubin II
direct bilirubin (DB) I | At baseline
  Blood concentration of direct bilirubin I
DB II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of direct bilirubin II
gamma-glutamyltransferase (GGTP) I | At baseline
  Blood concentration of gamma-glutamyltransferase I
GGTP II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of gamma-glutamyltransferase II
total cholesterol (TCH) I | At baseline
  Blood concentration of total cholesterol I
TCH II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of total cholesterol II
low density lipoprotein (LDL) I | At baseline
  Blood concentration of low density lipoprotein I
LDL II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of low density lipoprotein II
high density lipoprotein (HDL) I | At baseline
  Blood concentration of high density lipoprotein I
HDL II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of high density lipoprotein II
triglycerides (TG) I | At baseline
  Blood concentration of triglycerides I
TG II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of triglycerides II
apolipoprotein A (ApoA) I | At baseline
  Blood concentration of apolipoprotein A I
ApoA II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of apolipoprotein A II
insulin (INS) I | At baseline
  Blood concentration of insulin I
INS II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of insulin II
glucose (GLU) I | At baseline
  Blood concentration of glucose I
GLU II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of glucose II
creatinine (CREA) I | At baseline
  Blood concentration of creatinine I
CREA II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of creatinine II
C-reactive protein (CRP) I | At baseline
  Blood concentration of C-reactive protein I
CRP II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of C-reactive protein II
adropin (ADR) I | At baseline
  Blood concentration of adropin I
ADR II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of adropin II
neopterin (NEOPT) I | At baseline
  Blood concentration of neopterin I
NEOPT II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of neopterin II
N-terminal natriuretic propeptide type B (NTpro-BNP) I | At baseline
  Blood concentration of N-terminal natriuretic propeptide type B I
NTpro-BNP II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of N-terminal natriuretic propeptide type B II
magnesium (Mg) I | At baseline
  Blood concentration of magnesium I
Mg II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of magnesium II
homocysteine (Hcy) I | At baseline
  Blood concentration of homocysteine I
Hcy II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of homocysteine II
troponin (TROP) I | At baseline
  Blood concentration of troponin I
TROP II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of troponin II
interleukin 6 (IL6) I | At baseline
  Blood concentration of interleukin 6 I
IL6 II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of interleukin 6 II
tumor necrosis factor (TNF) I | At baseline
  Blood concentration of tumor necrosis factor I
TNF II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of tumor necrosis factor II
vascular endothelial growth factor (VEGF) I | At baseline
  Blood concentration of vascular endothelial growth factor I
VEGF II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of vascular endothelial growth factor II
leptin (LPT) I | At baseline
  Blood concentration of leptin I
LPT II | After intervention completion- an average of 2 weeks from baseline
  Blood concentration of leptin II
VEGF polymorphism | At baseline
  Polymorphism of the VEGF gene
Urine concentration of magnesium (U-Mg) I | At baseline
  Urine concentration of magnesium I
U-Mg II | After intervention completion- an average of 2 weeks from baseline
  Urine concentration of magnesium II
Hair content of magnesium (H-Mg) I | At baseline
  Hair content of magnesium I
H-Mg II | After intervention completion- an average of 2 weeks from baseline
  Hair content of magnesium II

CONTACTS AND LOCATIONS:
Overall Officials: Damian Skrypnik, MD; PhD, Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Department of Treatment of Obesity, Metabolic Disorders and Clinical Dietetics, Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No
The decision of individual participant data (IPD) sharing may be changed in the future.

REFERENCES:
- [Derived] Skrypnik D, Skrypnik K, Granell JC, Woszczyk D, Suliburska J. Cardiac rehabilitation influences serum myokine levels in patients after acute coronary syndrome: the randomised CARDIO-REH study. Sci Rep. 2025 Nov 6;15(1):38951. doi: 10.1038/s41598-025-22897-0. PMID 41198895
- [Derived] Skrypnik D, Skrypnik K, Suliburska J, Bogdanski P. Cardiac rehabilitation may influence leptin and VEGF A crosstalk in patients after acute coronary syndrome. Sci Rep. 2022 Jul 12;12(1):11825. doi: 10.1038/s41598-022-16053-1. PMID 35821400